CLINICAL TRIAL: NCT03219723
Title: Drug Use Surveillance of Takecab Tablets "Supplement to Helicobacter Pylori Eradication"
Brief Title: Drug Use Surveillance of Takecab for "Supplement to Helicobacter Pylori Eradication"
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Vonoprazan-5002; JapicCTI-153003 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2017-07-09; First posted 2017-07-17 (Actual); Results first posted 2019-03-22 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2018-12

CONDITIONS: Gastric/Duodenal Ulcer, Gastric MALT Lymphoma, Idiopathic Thrombocytopenic Purpura, or H. Pylori Gastritis, and Other
MeSH Terms: conditions — Duodenal Ulcer; Purpura, Thrombocytopenic, Idiopathic | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Clarithromycin; Metronidazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vonoprazan 20 mg: For adults, the following three-drug regimen will be administered orally at the same time twice daily for 7 days: 20 mg dose of vonoprazan, 750 mg (potency) dose of amoxicillin hydrate, and 200 mg (potency) dose of clarithromycin. The dose of clarithromycin may be increased as clinically warranted. However, dosage should not exceed 400 mg (potency)/dose twice daily. If H. pylori eradication with a three-drug regimen comprising vonoprazan or proton pump inhibitor + amoxicillin hydrate + clarithromycin has been unsuccessful, as an alternative treatment, the following three drugs will be administered orally twice daily for 7 days to adults: 20 mg dose of vonoprazan, 750 mg (potency) dose of amoxicillin hydrate, and 250 mg dose of metronidazole. Participants will receive interventions as part of routine medical care.
  Interventions: Drug: Vonoprazan; Drug: Amoxicillin hydrate; Drug: Clarithromycin; Drug: Metronidazole

INTERVENTIONS:
Drug: Vonoprazan — Vonoprazan tablets
  Other Names: Takecab tablets; TAK-438
Drug: Amoxicillin hydrate — Amoxicillin hydrate (potency)
Drug: Clarithromycin — Clarithromycin (potency)
Drug: Metronidazole — Metronidazole

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy on participants receiving first-line eradication and second-line eradication including vonoprazan (Takecab) tablets (triple therapy) in the routine clinical setting.

DETAILED DESCRIPTION:
The drug being tested in this study is called Vonoprazan (Takecab). Vonoprazan is being tested to treat people who have gastric ulcer, duodenal ulcer, gastric mucosa-associated lymphoid tissue (MALT) lymphoma, idiopathic thrombocytopenic purpura, stomach following endoscopic treatment of early gastric cancer, or H. pylori gastritis. This study will look at the presence or absence of new concerns regarding the safety of triple therapy with Vonoprazan tablets, amoxicillin, and clarithromycin (first-line eradication) and triple therapy with Vonoprazan tablets, amoxicillin, and metronidazole (second-line eradication) for supplemental Helicobacter pylori (H. pylori) eradication in the routine clinical setting. The study will enroll approximately 500 patients.

First-line eradication

* Vonoprazan 20 mg / Proton pump inhibitor
* Amoxicillin hydrate 750 mg
* Clarithromycin 200 mg

If H. pylori eradication with a three-drug regimen comprising vonoprazan or proton pump inhibitor + amoxicillin hydrate + clarithromycin has been unsuccessful.

Second-line eradication

* Vonoprazan 20 mg
* Amoxicillin hydrate 750 mg
* metronidazole 250 mg

This multi-center trial will be conducted in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Participants receiving H. pylori eradication treatment for the first time
* Participants for whom H. pylori eradication with Takecab tablets or proton pump inhibitor + amoxicillin + clarithromycin was found unsuccessful and who will receive eradication treatment with amoxicillin and metronidazole

Exclusion Criteria:

* Participants with previous history of hypersensitivity to ingredients in Takecab tablets
* Participants taking atazanavir sulfate or rilpivirine hydrochloride

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of participants receiving first-line eradication and second-line eradication including Takecab tablets (triple therapy) in the routine medical care.
Sampling Method: Probability Sample
Enrollment: 560 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda Selected Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 58 investigative sites in Japan, from 01 September 2015 to 30 April 2017.
Pre-assignment Details: Participants with a historical diagnosis of gastric/duodenal ulcer, idiopathic thrombocytopenic purpura, stomach following endoscopic treatment of early gastric cancer, or H. pylori gastritis were enrolled to receive interventions as part of routine medical care. However, participants with gastric MALT lymphoma were not enrolled in the survey.
Groups:
- Vonoprazan 20 mg: For adults, the following three-drug regimen was administered orally at the same time twice daily for 7 days: 20 mg dose of vonoprazan, 750 mg (potency) dose of amoxicillin hydrate, and 200 mg (potency) dose of clarithromycin. The dose of clarithromycin allowed to be increased as clinically warranted. However, dosage was not to exceed 400 mg (potency)/ dose twice daily. If H. pylori eradication with a three-drug regimen comprising vonoprazan or proton pump inhibitor + amoxicillin hydrate + clarithromycin had been unsuccessful, as an alternative treatment, the following three-drug regimen was administered orally twice daily for 7 days to adults: 20 mg dose of vonoprazan, 750 mg (potency) dose of amoxicillin hydrate, and 250 mg dose of metronidazole. Participants received interventions as part of routine medical care.
Period: Overall Study
Arm/Group | Vonoprazan 20 mg
Started | 560
Completed | 550
Not Completed | 10
Not completed — Case Report Forms Uncollected | 6
Not completed — Protocol Deviation | 4

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set; The safety analysis set was defined as all participants who completed the study.
Arm/Group | Vonoprazan 20 mg
Number analyzed (Participants) | 550
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.7 (13.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 293
  Male | 257
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  Japan | 550
Trial Indications [Count of Participants; unit: Participants] — EGC=Early Gastric Cancer. Participants could be counted in more than 1 category (including duplicates).
  Participants
    Gastric Ulcer | 50
    Duodenal Ulcer | 31
    Idiopathic Thrombocytopenic Purpura | 12
    Stomach Following Endoscopic Treatment of EGC | 12
    H. Pylori Gastritis | 476
Healthcare Category [Count of Participants; unit: Participants] — Participants were categorized as outpatient, inpatient.
  Participants
    Outpatient | 546
    Inpatient | 4
Predisposition to Hypersensitivity [Count of Participants; unit: Participants] — The baseline characteristic was analyzed in participants who had a liability or tendency to suffer from hypersensitivity.
  Participants
    Had Predisposition to Hypersensitivity | 16
    Had No Predisposition to Hypersensitivity | 518
    Unknown | 16
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had Presence of Medical Complications | 232
    Had No Presence of Medical Complications | 318
Pre-Therapy of H. Pylori Eradication before Study [Count of Participants; unit: Participants] — Population: Reported data was the number of participants who H. pylori eradication has been unsuccessful in pre-treatment by Vonoprazan or PPI, AMPC and CAM before this study (totally 48 participants).
  Participants
    number analyzed (Participants) | 48
    PPI + AMPC + CAM 400 mg | 7
    PPI + AMPC + CAM 800 mg | 27
    Vonoprazan + AMPC + CAM 400 mg | 4
    Vonoprazan + AMPC + CAM 800 mg | 7
    Unknown | 3
Height [Mean (Standard Deviation); unit: Centimeters (cm)] — Population: The number analyzed is the number of participants with data available for analysis.
  Centimeters (cm)
    number analyzed (Participants) | 306
    (all) | 160.62 (9.148)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] — Population: The number analyzed is the number of participants with data available for analysis.
  Kilograms (kg)
    number analyzed (Participants) | 318
    (all) | 59.63 (11.377)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight (kg)/[height (m)^2] Population: The number analyzed is the number of participants with data available for analysis.
  kg/m^2
    number analyzed (Participants) | 304
    (all) | 23.03 (3.481)
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 266
  Current Smoker | 67
  Ex-Smoker | 68
  Unknown | 149
Drinking Habits [Count of Participants; unit: Participants] — Participants who answered Yes or No for a question "Drink Alcohol Almost Every Day?" were reported.
  Participants
    Yes | 118
    No | 302
    Unknown | 130
Diagnostic Test for H. Pylori Infection [Count of Participants; unit: Participants] — Participants could be counted in more than 1 category (including duplicates).
  Participants
    Rapid Urease Test | 103
    Microscopy | 43
    Culture Method | 26
    Urea Breath Test | 167
    Anti-H. Pylori Antibody Test | 209
    Stool H. Pylori Antigen Test | 12
Treatment [Count of Participants; unit: Participants]
  First-Line Eradication | 502
  Second-Line Eradication | 48

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Had One or More Adverse Drug Reactions
Description: Adverse drug reaction refers to adverse events related to administered drug. Timeframe was defined as duration of triple therapy (7 days) and up to the time of determination of H. pylori eradication after triple therapy (approximately 2 months as maximum duration).
Time Frame: Up to 7 days and 2 months
Population: Safety Analysis Set; The safety analysis set was defined as all participants who completed the study.
Measure: Number; unit: Percentage of Participants
Arm/Group | Vonoprazan 20 mg
Number analyzed (Participants) | 550
Percentage of Participants | 3.09

2. Secondary Outcome: H. Pylori Eradication Rate
Description: In participants who were determined as achieving H. pylori eradication, the percentage of participants negative for H. pylori (eradication rates) was tabulated by first-line eradication and second-line eradication. Timeframe was defined as duration of triple therapy (7 days) and up to the time of determination of H. pylori eradication after triple therapy (approximately 2 months as maximum duration).
Time Frame: 7 days + 2 months
Population: Efficacy assessment population; The efficacy assessment population was defined as participants who completed the study and had efficacy data at baseline and post-baseline time points available.
Measure: Number (95% Confidence Interval); unit: Percent
Arm/Group | Vonoprazan 20 mg
Number analyzed (Participants) | 550
Percent
  First-Line Eradication: number analyzed (Participants) | 469
  First-Line Eradication | 91.24 [88.30 to 93.64]
  Second-Line Eradication: number analyzed (Participants) | 44
  Second-Line Eradication | 95.45 [84.53 to 99.44]

ADVERSE EVENTS:
Time Frame: Up to 7days and 2 months
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Vonoprazan 20 mg
All-Cause Mortality (participants affected / at risk) | 0/550
Serious Adverse Events (participants affected / at risk) | 0/550
Other Adverse Events (participants affected / at risk) | 22/550
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vonoprazan 20 mg (N=550)
Influenza (Infections and infestations) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 3
Hypogeusia (Nervous system disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 4
Faeces hard (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 1
Paraesthesia oral (Gastrointestinal disorders) | 1
Faeces soft (Gastrointestinal disorders) | 2
Liver disorder (Hepatobiliary disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1
Malaise (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT03219723/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-08): https://cdn.clinicaltrials.gov/large-docs/23/NCT03219723/SAP_001.pdf